CLINICAL TRIAL: NCT02518152
Title: Efficacy Of Platelet Rich Fibrin With 1% Alendronate For Treatment Of Intrabony Defects In Chronic Periodontitis: A Randomized Controlled Clinical Trial
Brief Title: Platelet Rich Fibrin+1% Alendronate in Treatment of Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Dr. A R Pradeep, Professor, Government Dental College and Research Institute, Bangalore, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2013-2014N
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Scaling and Root Planing (SRP) with Open flap debridement (OFD) alone for treating periodontal defect
  Interventions: Procedure: Open flap debridement (OFD)
- Group 2 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF) for treating periodontal defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)
- Group 3 (Active Comparator): SRP with Open flap debridement (OFD) with Platelet rich fibrin (PRF)+1% Alendronate for treating periodontal defect
  Interventions: Procedure: OFD with Platelet rich fibrin (PRF)+1% Alendronate

INTERVENTIONS:
Procedure: Open flap debridement (OFD) — Oral prophylaxis followed by Open flap debridement (OFD)
  Arms: Group 1
Procedure: OFD with Platelet rich fibrin (PRF) — Oral prophylaxis followed by Open flap debridement (OFD) with Platelet rich fibrin (PRF) placement into the bone defect
  Arms: Group 2
Procedure: OFD with Platelet rich fibrin (PRF)+1% Alendronate — Oral prophylaxis followed by Open flap debridement (OFD) with Platelet rich fibrin (PRF)+1% Alendronate placement into the bone defect
  Arms: Group 3

SUMMARY:
The present study is designed to evaluate the combined efficacy of Platelet Rich Fibrin (PRF) and 1% Alendronate (ALN) with open flap debridement (OFD) in treatment of intrabony defects in chronic periodontitis patients.

DETAILED DESCRIPTION:
Background: Platelet-rich fibrin (PRF) is a second-generation platelet concentrate, act as reservoirs of growth factors and cytokines which are the key factors for regeneration of the bone and maturation of the soft tissue. Alendronate (ALN), a potent member of bisphosphonate group is known to promote tissue regeneration by inhibiting osteoclastic bone resorption and promoting osteoblastogenesis. The present study was designed to evaluate the combined efficacy of PRF and 1% ALN with open flap debridement (OFD) in treatment of intrabony defects in chronic periodontitis patients.

Methods: Ninety patients with single defects were categorized into three groups: OFD alone, OFD with PRF,OFD with PRF+1% ALN. Clinical parameters; site specific plaque index (PI), modified sulcus bleeding index (mSBI), probing depth (PD), clinical attachment level (CAL) and gingival marginal level (GML) were recorded at baseline before surgery and 9 months post-operatively. Percentage radiographic intra-bony defect depth reduction (IBD) was evaluated at baseline and 9 months.

ELIGIBILITY:
Inclusion criteria

* Presence of 3-wall IBD ≥3 mm deep (distance between alveolar crest and base of the defect on an Intra-oral Periapical Radiograph [IOPA]) along with an interproximal probing depth (PD) ≥5 mm after phase I therapy (scaling and root planing[SRP]) in asymptomatic teeth.

Exclusion Criteria:

* Aggressive Periodontitis patients;
* Systemic conditions known to affect the periodontal status;
* medications known to affect the outcomes of periodontal therapy;
* Hematological disorders and insufficient platelet count (<200,000/mm3);
* Pregnancy/lactation;
* Smoking and tobacco use in any form
* Immunocompromised individuals.
* Those having unacceptable oral hygiene (plaque index27 [PI] >1.5) after reevaluation of Phase I therapy .
* Teeth with furcation involvement, non-vital teeth, carious teeth indicated for restorations and mobility of at least grade II were also excluded.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
defect depth reduction (%) | Change from baseline to 9 months
  assessed in percentage

SECONDARY OUTCOMES:
probing depth (mm) | Change from baseline to 9 months
  measured in mm
clinical attachment level (mm) | Change from baseline to 9 months
  measured in mm
gingival marginal level (mm) | Change from baseline to 9 months
  measured in mm
modified sulcus bleeding index | Change from baseline to 9 months
  scale from 0-3
plaque index | Change from baseline to 9 months
  scale from 0-3

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India